Grant Number: 1R01HD102545-01A4

ID: 750932-25 NCT05284006

Principal Investigator(s): Shunji Tomatsu, MD, PhD

Project Title: Non-invasive functional assessment and pathogenesis of Morquio A

Date of Document: March 11, 2025

#### **Accomplishments**

The long-term goal of this research proposal is to better understand the natural history of MPS IVA in terms of clinical progression and objective outcome measures. The unique aspect of our research is the establishment of innovative non-invasive assessments to evaluate the clinical severity, disease stage, and therapeutic efficacy of skeletal dysplasia. Our central hypothesis is that these assessments, when combined into a disease severity scoring system, can effectively characterize MPS IVA and assess the benefits of therapeutic interventions.

Aim 1. Conduct multidisciplinary and detailed non-invasive assessments in Morquio A patients. Our working hypothesis is that longitudinal non-invasive tests demonstrate accurate prognostic and predictive evaluation of skeletal dysplasia and can be carried out across a broad patient group, including patients who are young, wheelchair-bound, and post-surgical.

**Aim 2. Identify potential surrogate biomarkers of skeletal dysplasia.** Our working hypothesis is that biochemical biomarkers correlate with disease stage, clinical severity, and non-invasive clinical assessments. These biomarkers should, therefore, serve as prognostic and/or predictive biomarkers of therapeutic response.

# 1. Major activities Aims 1 and 2.

#### a. Team structure:

As outlined in the grant proposal, we assembled a dedicated and expert study team on May 1, 2021 (Fig. 1), demonstrating our unwavering commitment to the project.

-Monthly-based videoconferences between PI and investigators or board members from 6 Morquio A families have been set up since May 2021 to discuss the recruitment process, research plan, summary, and report on the project.



Figure 1. Structure of Study Team of Natural History

- b. Recruitment: During the COVID-19 pandemic, the recruitment process was significantly impacted, leading to delays due to limited access to the families and the hospital, and the requirement of vaccines to visit the hospital. Despite these challenges, sixty-two patients have consented to the study (Figures 2 and 3). Sixty patients have completed first visits, and thirty-eight have completed second visits. Twenty-one surgical specimens have been collected from participants. See the table below.
- **c. Data Collection:** This study includes 15 major assessments: clinical assessment procedures; anthropometric measurements; activity of daily living and quality-of-life questionnaires; gait kinematics and kinetics analysis; pulmonary function tests (PFT); skeletal radiographs and dual-energy x-ray absorptiometry (DXA); MRI in cervical spine, temporal bones, and hip; computed tomography angiography (CTA) for tracheal obstruction; CT for temporal bones; anesthetic encounters; joint mobility; hearing function; biochemical analyses; and pathological analyses.
  - In Aim 1, we have conducted all tests except for biochemical analysis. In Aim 2, we have analyzed some portions of data and will submit it to the articles,

### **Planned**

| Ethnic Categories | | | | | |
|---|---|---|---|---|---|
| | | oanic or<br>ino | Hispanic | Total | |
| Racial Categories | Female | Male | Female | Male | |
| American Indian/Alaska<br>Native | 0 | 0 | 0 | 0 | 0 |
| Asian | 3 | 3 | 0 | 0 | 6 |
| Native Hawaiian or Other<br>Pacific Islander | 0 | 0 | 0 | 0 | 0 |
| Black or African American | 4 | 4 | 0 | 0 | 8 |
| White | 20 | 20 | 0 | 0 | 40 |
| More than One Race | 0 | 0 | 3 | 3 | 6 |
| Total | 27 | 27 | 3 | 3 | 60 |

**Cumulative (Actual)** 

| Cumulative (Actual) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Ethnic Categories | | | | | | | | | | |
| | Not I | Hispanic or | Latino | His | Hispanic or Latino | | | Unknown/Not Reported | | |
| | | | Unknown/ | | | Unknown/ | | | Unknown/ | |
| | | | Not | | | Not | | | Not | |
| Racial Categories | Female | Male | Reported | Female | Male | Reported | Female | Male | Reported | |
| American Indian/Alaska Native | 1 | 1 | 0 | 0 | | 0 | 0 | 0 | 0 | 2 |
| Asian | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 |
| Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | 0 |
| Black or African American | 1 | 2 | 0 | 0 | | 0 | 0 | 0 | 0 | 3 |
| White | 26 | 14 | | 4 | 2 | | | | | 46 |
| More than One Race | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 |
| Unknown or Not Reported | 2 | 1 | | 1 | 1 | | | 1 | | 6 |
| Total | 29 | 18 | 0 | 6 | 4 | 0 | 0 | 1 | 0 | 66 |

| Age Enrollment Report | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Unknown/ | |
| | | | | | | | | | | Not | |
| Age Categories | 0-1 | 25 | 612 | 1317 | 1825 | 2645 | 4664 | 65-75 | 76+ | Reported | Total |
| Total | 2 | 13 | 19 | 5 | 12 | 14 | 1 | * | * | * | 66 |

<sup>•</sup>Currently Consented/Enrolled: 66

## d. Summary of Demographics

<sup>•</sup>Withdrawn: 11

<sup>•</sup>First visits: 64 complete, 2 scheduling

<sup>•</sup>Second Visits: 49 complete, 0 scheduling, 6 missed visits

<sup>•</sup>Third Visits: 4 complete, 17 scheduling

<sup>•</sup>Surgical Samples Collected: 25







Figure 2. Geographic maps (Global and US only)



Figure 3. Gender and Age



Figure 4. Racial Background



Figure 5. Race: Morquio Study vs. US Population



Figure 6. Ethnic Demographics



Figure 7. Ethnicity: Morquio A Study vs. US Population

#### 2. Specific objectives

Establishment of innovative non-invasive assessments to evaluate the clinical severity, disease stage, and therapeutic efficacy of skeletal dysplasia.

Aim 1. Conduct multidisciplinary and detailed non-invasive assessments in Morquio A patients. Our working hypothesis is that longitudinal non-invasive tests demonstrate accurate prognostic and predictive assessment of skeletal dysplasia and can be carried out across a broad patient group, including patients who are young, wheelchair-bound, and post-surgical.

**Aim 2. Identify potential surrogate biomarkers of skeletal dysplasia.** Our working hypothesis is that biochemical biomarkers correlate with disease stage, clinical severity, and non-invasive clinical assessments. These biomarkers should, therefore, serve as prognostic and/or predictive biomarkers of therapeutic response.

3. Significant results (including) major findings, developments, or conclusions (both positive and negative)

Aims 1 and 2.

- We have completed the first visits for 64 patients, the second for 49 patients, and the third for four patients, 17 scheduling in the problematic situation of COVID-19 after confirming the safety and feasibility of the families. 25 Surgical Samples were Collected.
  - We recruited the patients, including 5 international patients. We assume 15 % of the MPS IVA patients in the USA participated in this program if around 400 MPS IVA patients are present. This is very significant in terms of the number of patients. Also, the demographics of the participants are similar to the USA ethnic population pattern, which MPS IVA incidence happens in diverse populations.
- 2. Until now, no patient has had any discomfort or incapability with the proposed tests, which matches our hypothesis that all non-invasive tests are feasible for patients without age or physical handicap. Our non-invasive tests are feasible and acceptable to the majority of patients compared to endurance tests, which include a 6 min walk test and a 3 min climb-up test. This is one of our major goals and a significant result.
- 3. We found that NTproCNP is currently the most promising biomarker during the study. We plan to measure this biomarker continuously in human blood and urine to identify the correlation between skeletal dysplasia and NTproCNP level. In addition, we are exploring the potential of CNP as a therapeutic agent on the MPS IVA animal models. The discovery of NTproCNP is significant as a potential surrogate biomarker and can be used for the future clinical trial.
- 4. Based on the natural history program activity and data, our project is selected for the clinical trial the Foundation for the National Institutes of Health (FINH) <u>Accelerating Medicines Partnership® Bespoke Gene Therapy Consortium</u> (AMP® BGTC), which is public-private partnership between the NIH, U.S. Food and Drug Administration (FDA), biopharmaceutical and life sciences companies, and non-profit and other organizations to develop and deliver bespoke (i.e., customized) gene therapies to treat patients with rare diseases. <u>AMP® BGTC</u> aims to accelerate the development and approval of gene therapies for eight rare diseases, including Morquio A Syndrome. This is a very significant result for the entire Morquio Community, Researchers, and
  - We have a schedule of the clinical trial for Morquio A in 2027 using AAV gene therapy. The current data will be used for the baseline data of the clinical trial.
- 5. Because of COVID-19, we have delayed collecting data, which is a serious issue to have longitudinal data (4 visits).

#### 4. Key outcomes or other achievements

#### Aims 1 and 2.

**Identify potential surrogate biomarkers of skeletal dysplasia.** Our working hypothesis is that biochemical biomarkers correlate with disease stage, clinical severity, and non-invasive clinical assessments. These biomarkers should, therefore, serve as prognostic and/or predictive biomarkers of therapeutic response. We collected urine and blood samples from patients who visited the hospital on the first, second, and third visits.

#### Materials and methods

#### **Subjects**

MPS IVA patients

MPS IVA patients commuting to Nemours Children's Hospital in Delaware have participated. Written informed consent was obtained before any study procedures were conducted.

#### **Controls**

Residual serum from various patients without skeletal dysplasia at Shimane University Hospital was frozen after biochemical analysis and then sent to our laboratory as control samples for this research. The patients ranged in age from 0 day to 16 years. Blood samples were also collected from 7 healthy adults working in this laboratory, and both plasma and serum were stored. Written informed consent was obtained from them.

#### a. Collagen type I

Human Collagen Type I (COL1) ELISA Kit (Cat# EKU03297-96T, BIOMATIK, Kitchener, Canada) was used to measure the concentration of collagen type I in patient plasma and control serum and control plasma according to the manufacturer's instructions.

#### b. Collagen type II

Human Collagen Type II, Col II ELISA Kit (Cat# EKC40379, BIOMATIK, Kitchener, Canada) was used to measure the concentration of collagen type II in patient plasma and control serum and control plasma according to the manufacturer's instructions.

#### c. Collagen type X

Human Collagen X ELISA Kit (Colorimetric) (Cat# NBP2-75826, Novus Biologicals, Centennial, Colorado, USA) was used to measure the concentration of collagen type X in patient plasma and control serum and control plasma according to the manufacturer's instructions.

#### d. NT-proCNP

NT-proCNP ELISA kit (Cat# BI-20812, BIOMEDICA, Vienna, Austria) was used to measure the concentration of amino-terminal pro C type natriuretic peptide (NT-proCNP) in patient plasma and control serum and control plasma according to the manufacturer's instructions.

#### e. Anti-rhGALNS IgG

Enzyme-Linked Immunosorbent Assay (ELISA) was used to measure the concentration of anti-rhGALNS IgG in each sample.

#### f. Anti-AAV8 IgG and Anti-AAV9 IgG

The ELISA method [1] was used with modifications to detect these antibodies.

#### g. Genotype

The genomic DNA of each patient was extracted from frozen WBC, and then all 14 exons in the GALNS gene were PCR-amplified and sequenced by the Sanger method to detect pathogenic mutations.

### h. Glycosaminoglycans (GAG) analysis by LC-MS/MS

**Control serum and urine:** We obtained serum and urine from various patients without skeletal dysplasia at Shimane University Hospital. Control serum ages 5-18 years and urine 5-33 years

# Results (outcomes) Collagen type I and II



Figure 1. Collagen type I (A) and II (B) levels in patients and controls. Both vertical axes are presented on a base-2 logarithmic scale.

#### a. Collagen type I

We found a statistically significant increase in collagen type I in patients older than 20 (**Table 1**, **Figure 1 (A)**). **Table 1**. **Comparison of collagen type I levels in 5 age groups.** 

| Age | No. | Mean | SD | Maximum | Minimum | Mean<br>age | p-value |
|---|---|---|---|---|---|---|---|
| Control | | | | | | | |
| ≤ 1 y | 1 | 2803.4 | 0 | 2803.4 | 2803.4 | 0.25 | |
| >1, ≤ 5 y | 4 | 2715.5 | 2400.5 | 6397.5 | 329.6 | 2.51 | |
| >5, ≤ 10 y | 6 | 1019.0 | 481.2 | 2039.0 | 566.0 | 7.19 | |
| >10, ≤ 15 y | 5 | 1572.0 | 2123.6 | 5734.8 | 32.9 | 11.98 | |
| > 15, ≤ 20<br>y | 1 | 996.1 | 0 | 996.1 | 996.1 | 15.99 | |
| >20 y | 7 | 76.6 | 18.6 | 106.3 | 49.3 | 39.57 | |
| MPS IVA | | | | | | | |
| >1, ≤ 5 y | 8 | 1022.4 | 681.8 | 2654.1 | 490.7 | 3.05 | 0.31 |
| >5, ≤ 10 y | 24 | 679.4 | 469.3 | 1630.2 | 50.3 | 7.38 | 0.19 |
| >10, ≤ 15 y | 14 | 752.4 | 398.1 | 1722.0 | 381.2 | 12.52 | 0.48 |
| > 15, ≤ 20<br>y | 11 | 323.9 | 314.8 | 1161.6 | 67.0 | 17.70 | N/A |
| >20 y | 41 | 125.7 | 92.1 | 383.0 | 24.5 | 33.35 | 0.0046 |

#### b. Collagen type II

We found a statistically significant increase in collagen type II in patients in two age groups, between 5 and 10 years and over 20 years (**Table 2**, **Figure 1** (**B**)). We calculated the partial correlation coefficient between collagen type II and NT-proCNP, controlling for age using the entire age group. There was almost no correlation (r = 0.042, p = 0.69).

Table 2. Comparison of collagen type II levels in 5 age groups.

| Age | No. | Mean | SD | Maximum | Minimum | Mean age | p-value |
|---|---|---|---|---|---|---|---|
| Control | | | | | | | |
| >1, ≤ 5 y | 18 | 129.03 | 92.41 | 324.99 | 11.70 | 2.68 | |
| >5, ≤ 10 y | 12 | 113.70 | 53.62 | 231.40 | 36.66 | 6.97 | |
| >10, ≤ 15 y | 7 | 85.64 | 78.26 | 253.57 | 16.66 | 12.21 | |
| > 15, ≤ 20 y | 2 | 43.85 | 30.83 | 74.68 | 13.02 | 16.50 | |
| >20 y | 7 | 35.72 | 22.85 | 76.23 | 10.51 | 39.57 | |
| MPS IVA | | | | | | | |
| >1, ≤ 5 y | 7 | 105.80 | 74.15 | 240.58 | 29.44 | 3.23 | 0.55 |
| >5, ≤ 10 y | 21 | 234.54 | 233.64 | 885.55 | 15.93 | 7.30 | 0.037 |
| >10, ≤ 15 y | 14 | 70.07 | 59.39 | 208.32 | 17.03 | 12.52 | 0.67 |
| > 15, ≤ 20 y | 11 | 131.71 | 181.03 | 534.18 | 12.77 | 17.70 | 0.21 |
| >20 y | 40 | 90.71 | 105.27 | 438.58 | 6.10 | 33.54 | 0.0097 |

#### c. Collagen type X



**Figure 2.** Collagen type X levels in blood We did not find any significant difference or trend.

#### d. NT-proCNP



**Figure 3:** Correlation between age, NT-proCNP level in plasma, and height of patients with MPS IVA. Males and females are shown in the left and right figures, respectively. Round dots represent patients treated with enzyme replacement therapy (ERT). Triangle markers represent patients who were never treated with ERT. Square markers represent patients treated with hematopoietic stem cell transplantation (HSCT). Filled markers represent patients for whom height at blood sample collection was recorded. The color of each marker represents the z-score of each patient's height calculated based on the 2022 CDC growth chart. Black dotted lines show median, 5th and 95th percentiles for healthy controls [30]. When a patient has two data points, each data point is connected by a green dotted line.



Figure 4: The relationship between each patient's plasma NT-proCNP level, age, and subsequent height growth rate (height velocity): Height velocity was calculated from two sets of height data measured at different times, 7-20 months apart. Each dot represents the age of each patient at which the first height was measured (horizontal axis) and the corresponding later height velocity (vertical axis). Round dots represent patients who received ERT continuously until the second height data was obtained. The square dot represents a patient who had received HSCT. The triangular dot indicates a patient who never received ERT until his second height data was obtained. Larger round dots represent the attenuated phenotype, while smaller round dots represent the severe phenotype. Each dot is filled with a color corresponding to the plasma NT-proCNP level at the first height measurement. The light blue and pink lines show the 50th percentile for height velocity for male and female MPS IVA patients, respectively [29]. The gray dotted line shows the 50th percentile for height velocity for healthy males and females.

We revealed a significant increase of NT-proCNP in patients under 20 years (Welch's t-test,  $p = 2.67 \times 10^{-12}$ ). The increase was particularly evident just before the age of pubertal growth spurt in healthy subjects (**Fig. 3**). If we focus only on patients who have two data points at different ages before the age of pubertal growth spurt (all had received ERT during these two periods), 5 out of 10 boys and 2 out of 3 girls showed the increase in NT-proCNP level. This suggests that plasma NT-proCNP would not be a pharmacodynamic biomarker differing from urinary KS [10] before the age of pubertal growth spurt.

The concentration of NT-proCNP in plasma from patients under 20 years showed a negative correlation with age, and the correlation coefficient (r) was -0.612 ( $p = 7.44 \times 10^{-11}$ ). The Z-score of each patient's height showed a significant negative correlation with age, as current therapy is ineffective to prevent growth failure in MPS IVA (r = -0.703,  $p < 1.21 \times 10^{-6}$ ). We then calculated the partial correlation coefficient between NT-proCNP and z-score of height controlling for age, which is summarized in **Table 3 (below, partial correlation coefficient between NT-proCNP and z-score of height, controlling for age)**. We found a negative correlation after the age of 8 years.

| Age group | number<br>of<br>subjects | Partial correlation coefficient | p-value |
|---|---|---|---|
| ≤ 8 y | 20 | 0.19 | 0.4355 |
| >8, ≤ 13 y | 17 | -0.568 | 0.0217 |
| >13, ≤ 20 y | 15 | -0.837 | 1.865 × 10 <sup>-4</sup> |

In addition, for patients with more than two visits, height velocity was calculated from two sets of height data measured at different times, 7-20 months apart, as summarized in **Fig. 4**. These findings are consistent with the hypothesis in achondroplasia that elevated levels of CNP-related peptides are natural responses to disturbed bone growth [11, 12]. Further accumulation of data from MPS patients is essential

and urgent to determine the accurate correlation between NT-proCNP and skeletal symptoms, including height.





**Figure 5.** Anti-GALNS antibody levels in blood ERT is strongly associated with the elevation of anti-rhGALNS antibodies. One patient who received HSCT at 8 years had received ERT until HSCT.

# f. Anti-AAV8 IgG and Anti-AAV9 IgG Under investigation.

# g. Genotype: we have identified the following genotypes from participants.

| Patient | ì | onoty po | Height | Age | Geno | type | onowing g |
|---|---|---|---|---|---|---|---|
| ID<br>M01 | Sex<br>F | Race<br>White or Caucasian | (Z-score)<br>-6.34 | (year)<br>17.16 | Allele 1<br>c.740G>A (G247D) | Allele 2<br>c.901G>T (G301C) | T reatment<br>ERT |
| M02 | F | Chinese | -6.73 | 18.70 | c.953T>G(M318R) | c.1567T>G(X523EextX93) | ERT |
| | | | | 40.00 | | | |
| M03<br>M04 | F | White or Caucasian<br>White or Caucasian | | 24.62<br>42.12 | c.448delC (H150Tfs*3)<br>c.675dupC (F226Lfs*37) | c.651_652insG (K218Efs*45)<br>unknown | ERT<br>ERT |
| M05 | F | White or Caucasian | -9.93 | 43.51<br>18.35 | c.346G>A (G116S) | c.1156C>T (R386C) | ERT |
| | | | -9.76 | 19.78 | | | |
| M06 | F | White or Caucasian | -8.52 | 19.89<br>21.29 | c.346G>A (G116S) | c.1156C>T (R386C) | ERT |
| M07<br>M08 | M | White or Caucasian<br>White or Caucasian | no record | 32.25<br>8.00 | c.337A>T (I113F)<br>c.122T>A (M41K) | c.1171A>G (M391V)<br>c.122T>A (M41K) | No ERT for 2 years and 8 month<br>ERT |
| M10 | M | White or Caucasian | -6.09<br>1.22 | 9.03 | c.338T>C (I113T) | | Received HSCT 1 year ago<br>ERT |
| M10 | М | White or Caucasian | 1.01 | 10.82<br>12.37 | e.3381 ×C (11131) | c.1219A>C (N407H) | ERI |
| M11 | F | White or Caucasian | -5.36<br>-5.53 | 15.11 | c.421T>A (W141R) | unknown | ERT |
| M12 | F | White or Caucasian | | 26.65<br>28.15 | c.697G>A (D233N) | e.1034T>C (L345P) | No ERT for 4 years and 4 month |
| M13 | M | Black or African American | -7.52 | 13.13 | c.251C>A (A84E) | c.319G>A (A107T) | ERT |
| M14 | F | White or Caucasian | -6.75<br>-5.7 | 14.84 | c.740G>A (G247D) | unknown | ERT |
| M15 | M | White or Caucasian | -5.7<br>-2.39 | 17.83 | c.498delC (F167Lfs*32) | c.901G>T (G301C) | ERT |
| | | | -3.84 | 6.81 | | | |
| M16 | M | Filipino | -5.09<br>no record | 5.21<br>6.77 | c.228C>A (N76K) | c.1480A>G (p.M494V) | ERT |
| M19 | F | Black or African American | -6.49<br>-5.64 | 9.44<br>10.96 | c.245C>T (S82L) | unknown | ERT |
| M20 | F | White or Caucasian | -4.09 | 9.49 | c.498delC (F167Lfs*32) | c.1474G>A (A492T) | ERT |
| M21 | M | White or Caucasian | -3.53<br>-4.08 | 10.06<br>6.12 | c.651_652insG (K218Efs*45) | c.1159G>A (G387S) | ERT |
| M22 | M | White or Caucasian | -5.22<br>-5.45 | 7.55<br>8.34 | c.651_652insG (K218Efs*45) | c.1159G>A (G387S) | ERT |
| | | | -7.24 | 9.78 | | | |
| M25 | М | White or Caucasian | | 41.34 | c.155C>T (P52L) | c.337A>T (I113F) | Never received ERT |
| M26 | М | Filipino | -7.03<br>no record | 12.39<br>13.89 | c.93delC (N32Tfs*97) | c.946G>A (G316R) | ERT |
| M28 | F | Mixed | полесота | 31.20 | c.868G>A (G290S) | c.868G>A (G290S) | Never received ERT |
| M30 | F | Japanese and Caucasian<br>White or Caucasian | | 32.75<br>43.52 | c.121-12T>C | e.121-12T>C | ERT |
| M31 | M | Black or African American | -1.29<br>-1.11 | 9.86<br>11.44 | c.935C>G (T312S) | c.1520G>T (C507F) | ERT |
| M32 | F | White or Caucasian | | 45.50 | c.121-12T>C | e.121-12T>C | Never received ERT |
| M33 | F | White or Caucasian | | 47.03<br>29.94 | e.1012C>T (Q338X) | c.1171A>G (M391V) | Never received ERT |
| M34 | M | White or Caucasian | | 31.48<br>28.17 | c.121A>T (M41L) | c.121A>T (M41L) | ERT |
| | | | | 29.69 | | | |
| M35 | M | White or Caucasian | -6.86<br>-7.69 | 11.23<br>12.64 | c.139G>A (G47R) | c.1156C>T (R386C) | No ERT for 4 years |
| M36 | F | Asian Indian | | 25.72<br>27.27 | c.346G>A (GI16S) | c.346G>A (G116S) | ERT |
| M37 | M | Asian Indian | -10.12 | 19.01 | c.346G>A (GI16S) | c.346G>A (G116S) | ERT |
| M38 | F | White or Caucasian | -5.63 | 20.56<br>16.04 | c.1559G>A (W520X) | unknown | ERT |
| M39<br>M41 | F<br>M | White or Caucasian<br>White or Caucasian | -3.54 | 12.08<br>35.29 | c.1559G>A (W520X)<br>c.121A>T (M41L) | unknown<br>c.498delC (F167Lfs*32) | ERT<br>ERT |
| M42 | F | White or Caucasian | | 36.86<br>28.24 | c.860C>T (\$287L) | c.1055T>C (L352P) | ERT |
| | | | | 29.95 | | | |
| M43 | M | White or Caucasian | | 29.04<br>30.52 | c.121A>T (M41L) | c.901G>T (G301C) | ERT |
| M44 | F | White or Caucasian | | 24.28<br>25.85 | e.1171A>G (p.M391V) | c.502G>A (p.G168R) | ERT |
| M45 | F | White or Caucasian | | 61.08 | c.740G>A (G247D) | c.761A>G (Y254C) | Never received ERT |
| M46 | F | White or Caucasian | no record | 62.66 | c.167C>A (T56N) | c.502G>A (G168R) | ERT |
| M47 | F | Some other race | -5.54 | 8.40<br>24.33 | c.139G>A (G47R) | c.466T>C (F156L) | ERT |
| | | | | 25.78 | | | |
| M48 | F | White or Caucasian | -7.11<br>-7.66 | 13.23<br>14.68 | c.139G>A (G47R) | c.466T>C (F156L) | ERT |
| M49<br>M50 | M<br>F | White or Caucasian<br>White or Caucasian | -6.44<br>-3.33 | 7.68<br>5.65 | c.1156C>T (R386C)<br>c.451C>A (P151T) | c.1156C>T (R386C)<br>c.477G>A (W159X) | ERT<br>ERT |
| | | | -4.81 | 7.26 | | | |
| M51 | M | White or Caucasian | -0.9<br>-0.52 | 2.89<br>4.50 | c.451C>A (P151T) | c.477G>A (W159X) | ERT |
| M52 | F | Multiple Races | no record | 2.50<br>4.60 | c.651_652insG (K218Efs*45) | unknown | Received HSCT 11 months ago |
| | | | -2.54 | 6.21 | | | |
| M53 | F | Chinese | | 23.20<br>24.37 | e.1482+5G>C | c.1498G>T (G500C) | No ERT for 13 months<br>ERT |
| M54<br>M55 | F | White or Caucasian<br>White or Caucasian | -3.04 | 36.26<br>5.39 | not tested<br>c.1339G>C (D447H) | not tested<br>unknown | No ERT for 5 years and 9 month<br>ERT |
| | F | | -4.2 | 6.80 | | | |
| M56<br>M57 | М | White or Caucasian<br>White or Caucasian | -1.44<br>0.41 | 3.79<br>1.13 | c.740G>A (G247D)<br>c.740G>A(G247D) | c.1451C>A (P484H)<br>c.1451C>A (P484H) | Never received ERT Never received ERT |
| M58<br>M59 | M | White or Caucasian<br>White or Caucasian | -4.38<br>-4.14 | 6.78 | c.1012C>T (Q338X)<br>c.337A>T (p.I113F) | c.181C>G (R61G)<br>c.901G>T (p.G301C) | ERT<br>ERT |
| | F | Some other race | | 26.58 | c.901G>T (G301C) | c.1156C>T (R386C) | Never received ERT |
| M60 | _ | | | 22.72 | c.331C>T (Q111X) | c.1365-2A>G<br>c.1558T>C (W520R) | ERT<br>ERT |
| M60<br>M63<br>M64 | F | White or Caucasian<br>Black or African American | -3.74 | 5.64 | e.633+1G>C | C.15501 - C (11520K) | EKI |
| M63 | F | | -3.74<br>-2.9<br>-2.1 | 5.64<br>6.50<br>3.34 | c.633+1G>C | c.1558T>C (W520R)<br>unknown | ERT<br>ERT |
| M63<br>M64<br>M65 | F<br>M<br>M | Black or African American<br>Black or African American | -2.9 | 6.50 | | c.1558T>C (W520R) | ERT |

#### h. GAGs

The results of mono-sulfated KS, di-sulfated KS, KS ratio (the rate of di-sulfated KS among total KS), and C6S in urine and blood from patients are summarized in **Table 4** and **Figure 6**. For C6S, the number of available control samples was less than for KS, so the "number of samples" and "mean age" differed from KS in **Table 4**. Partial correlation coefficients controlling for age between z-score of height and each significant GAG (mono-sulfated and di-sulfated KS and urinary C6S) were calculated and summarized in **Table 5**.

Table 4. Summary of GAG levels in 5 age groups

| | _ | | | - | | | Number | |
|---|---|---|---|---|---|---|---|---|
| Age group | Number<br>of<br>samples | Mean<br>age | Mono-<br>sulfated KS | Di-sulfated KS | KS ratio (%) | C6S | of<br>sample<br>s | Mean<br>age |
| Control | (urine) | | | | | | | |
| >1, ≤ 5 y | 18 | 3.47 | 2128 ± 618 | 663 ± 263 | $23.4 \pm 4.6$ | N/A | 0 | N/A |
| >5, ≤ 10 y | 14 | 6.48 | 1380 ± 833 | 768 ± 439 | 36.8 ± 5.6 | 164.7 ±<br>129.7 | 14 | 6.48 |
| >10, ≤ 15 y | 15 | 12.75 | 971 ± 574 | 802 ± 413 | 46.5 ± 9.4 | 178.1 ±<br>104.1 | 15 | 12.75 |
| > 15, ≤ 20<br>y | 3 | 17 | 215 ± 96 | 271 ± 69 | 57.2 ± 4.9 | 83.3 ± 17.2 | 3 | 17 |
| >20 y | 6 | 37.92 | 157 ± 45 | 255 ± 283 | 48.7 ± 18.6 | 88.0 ± 19.8 | 3 | 31.03 |
| MPS IVA | (urine) | | | | | | | |
| >1, ≤ 5 y | 3 | 3.73 | 9202 ± 1563* | 20081 ± 2603** | 68.6 ± 3.6*** | 727 ± 282 | | |
| >5, ≤ 10 y | 23 | 7.24 | 9904 ±<br>5024*** | 18225 ±<br>9116*** | 63.9 ± 8.3*** | 633 ± 398*** | | |
| >10, ≤ 15 y | 15 | 12.36 | 8143 ±<br>10725* | 12343 ±<br>11876** | 65.1 ± 11.1*** | 465 ± 247*** | | |
| > 15, ≤ 20<br>y | 11 | 17.7 | 2340 ±<br>1178*** | 3091 ± 1509*** | 56.7 ± 8.0 | 289 ± 189** | | |
| >20 y | 39 | 33.56 | 2267 ±<br>1391*** | 4033 ± 2286*** | 64.4 ± 7.7 | 245 ± 131*** | | |
| Age group | Number<br>of<br>samples | Mean<br>age | Mono-<br>sulfated KS | Di-sulfated KS | KS ratio (%) | C6S | Number<br>of<br>sample<br>s | Mean<br>age |
| | of | | | Di-sulfated KS | KS ratio (%) | C6S | of<br>sample | |
| | of<br>samples | | | Di-sulfated KS<br>229 ± 40 | KS ratio (%)<br>17.4 ± 1.3 | C6S<br>5.15 ± 2.67 | of<br>sample | |
| Control | of<br>samples<br>(serum) | age | sulfated KS | | | | of<br>sample<br>s | age |
| <b>Control</b> >1, ≤ 5 y | of<br>samples<br>(serum)<br>4 | age<br>2 | sulfated KS<br>1095 ± 223 | 229 ± 40 | 17.4 ± 1.3 | 5.15 ± 2.67 | of<br>sample<br>s | age<br>2 |
| Control >1, ≤ 5 y >5, ≤ 10 y | of<br>samples<br>(serum)<br>4<br>17 | 2<br>7.18 | sulfated KS<br>1095 ± 223<br>660 ± 220 | 229 ± 40<br>197 ± 59 | 17.4 ± 1.3<br>23.3 ± 3.6 | 5.15 ± 2.67<br>2.34 ± 2.01 | of sample s | 2<br>7.18 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 | of samples (serum) 4 17 10 | 2<br>7.18<br>12.35 | sulfated KS<br>1095 ± 223<br>660 ± 220<br>545 ± 235 | 229 ± 40<br>197 ± 59<br>248 ± 88 | 17.4 ± 1.3<br>23.3 ± 3.6<br>32.3 ± 5.0 | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29 | of sample s 4 17 10 | 2<br>7.18<br>12.35 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 y >20 y | of samples (serum) 4 17 10 10 | 2<br>7.18<br>12.35<br>15.9 | sulfated KS<br>1095 ± 223<br>660 ± 220<br>545 ± 235<br>322 ± 123 | 229 ± 40<br>197 ± 59<br>248 ± 88<br>118 ± 73 | $17.4 \pm 1.3$ $23.3 \pm 3.6$ $32.3 \pm 5.0$ $27.8 \pm 14.7$ | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29<br>0.49 ± 0.06 | of sample s 4 17 10 2 | 2<br>7.18<br>12.35<br>17 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 y >20 y | of samples (serum) 4 17 10 10 15 | 2<br>7.18<br>12.35<br>15.9 | sulfated KS<br>1095 ± 223<br>660 ± 220<br>545 ± 235<br>322 ± 123 | 229 ± 40<br>197 ± 59<br>248 ± 88<br>118 ± 73 | $17.4 \pm 1.3$ $23.3 \pm 3.6$ $32.3 \pm 5.0$ $27.8 \pm 14.7$ | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29<br>0.49 ± 0.06 | of sample s 4 17 10 2 | 2<br>7.18<br>12.35<br>17 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 y >20 y MPS IVA | of samples (serum) 4 17 10 10 15 (plasma) | 2<br>7.18<br>12.35<br>15.9<br>42.2 | sulfated KS 1095 ± 223 660 ± 220 545 ± 235 322 ± 123 314 ± 109 | 229 ± 40<br>197 ± 59<br>248 ± 88<br>118 ± 73<br>86 ± 43 | $17.4 \pm 1.3$ $23.3 \pm 3.6$ $32.3 \pm 5.0$ $27.8 \pm 14.7$ $21.4 \pm 7.8$ | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29<br>0.49 ± 0.06<br>N/A | of sample s 4 17 10 2 | 2<br>7.18<br>12.35<br>17 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 y >20 y MPS IVA >1, ≤ 5 y | of samples (serum) 4 17 10 10 15 (plasma) 8 | 2<br>7.18<br>12.35<br>15.9<br>42.2 | sulfated KS 1095 ± 223 660 ± 220 545 ± 235 322 ± 123 314 ± 109 1805 ± 514* | 229 ± 40<br>197 ± 59<br>248 ± 88<br>118 ± 73<br>86 ± 43 | $17.4 \pm 1.3$ $23.3 \pm 3.6$ $32.3 \pm 5.0$ $27.8 \pm 14.7$ $21.4 \pm 7.8$ $33.7 \pm 4.1***$ | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29<br>0.49 ± 0.06<br>N/A | of sample s 4 17 10 2 | 2<br>7.18<br>12.35<br>17 |
| Control >1, ≤ 5 y >5, ≤ 10 y >10, ≤ 15 y >15, ≤ 20 y >20 y MPS IVA >1, ≤ 5 y >5, ≤ 10 y | of samples (serum) 4 17 10 10 15 (plasma) 8 22 | 2<br>7.18<br>12.35<br>15.9<br>42.2<br>3.13<br>7.33 | sulfated KS 1095 ± 223 660 ± 220 545 ± 235 322 ± 123 314 ± 109 1805 ± 514* 1556 ± 363*** | 229 ± 40<br>197 ± 59<br>248 ± 88<br>118 ± 73<br>86 ± 43<br>910 ± 229***<br>639 ± 227*** | $17.4 \pm 1.3$ $23.3 \pm 3.6$ $32.3 \pm 5.0$ $27.8 \pm 14.7$ $21.4 \pm 7.8$ $33.7 \pm 4.1***$ $28.7 \pm 6.0**$ | 5.15 ± 2.67<br>2.34 ± 2.01<br>2.81 ± 2.29<br>0.49 ± 0.06<br>N/A<br>1.97 ± 2.53<br>1.97 ± 3.88 | of sample s 4 17 10 2 | 2<br>7.18<br>12.35<br>17 |

<sup>\*</sup>p < 0.05, \*\*p < 0.01, \*\*\*p < 0.001



**Figure 6: Glycosaminoglycan levels in urine and blood.** Mono-sulfated KS, di-sulfated KS, KS ratio (di-sulfated KS to total KS), and C6S levels in urine and blood are summarized in scatter plots. The horizontal axes indicate the age (years) of each patient or control. For urinary mono-sulfated and di-sulfated KS levels, the vertical axes are shown on a base-10 logarithmic scale. Round red dots indicate patients who ever received ERT. Purple squares are indicated for patients who received HSCT. Gray triangles represent patients who never received ERT or HSCT. Green x marks represent controls. For blood samples, plasma samples were used for patients and serum for controls.

Table 5. The partial correlation coefficient (r) between each GAG and the z-score of height of patients under 20 years old, controlling for age

| | Number of subjects to calculate the <i>r</i> value | r | р |
|---|---|---|---|
| Urine di-sulfated KS | 49 | -0.484 | 0.00049 |
| Urine mono-sulfated KS | 49 | -0.42 | 0.00293 |
| Plasma di-sulfated KS | 50 | -0.041 | 0.777 |
| Plasma mono-sulfated KS | 50 | -0.181 | 0.213 |
| Urine C6S | 49 | -0.282 | 0.0517 |

#### Conclusions and plan

Collagen type I: This is not a significant biomarker for pediatric patients. Several papers reported that the expression level of mRNA encoding collagen type I increased in chondrocytes from human MPS IVA patients [13, 14]. Comprehensive proteomic analysis of 6-week-old mouse femurs also showed that collagen alpha-1 and 2 (Uniprot IDs: P11087 and Q01149) increased in MPS IVA [15]. Therefore, we predicted that patients would present with higher concentration levels than the control group. However, only adult patients showed such differences. On the contrary, other age groups showed lower concentration in patients, even though it was not statistically significant. Because human collagen type I has a molecular weight of approximately 300 kDa, much larger than NT-proCNP, and is surrounded by hydroxyapatite in bone [16–18]It could be pretty difficult for collagen type I to escape from bone and cartilage and enter the bloodstream compared to NT-proCNP, thereby preventing higher concentrations in the blood of patients. We should measure smaller peptides related to collagen type I.

**Collagen type II:** This is not a significant biomarker for pediatric patients. Blood procollagen II C-terminal propeptide (CPII) and/or urinary C-terminal telopeptide of type II collagen (CTX-II) are currently the two primary markers of type II collagen metabolism in osteoarthritis [19–21], joint injuries [22], and Kashin-Beck disease (KBD) [23]. CPII reflects the synthesis of type II collagen during cartilage repair and remodeling [24–26], while CTX-II is a marker of type II collagen breakdown, reflecting cartilage catabolism [21, 27]. We will consider focusing on these peptides related to collagen type II.

**Collagen type X:** No significant findings were obtained. Also, the kit I used (https://www.novusbio.com/products/collagen-x-elisa-kit\_nbp2-75826) is no longer manufactured. We will have to purchase other kits if we continue to measure this biomarker.

#### NTproCNP in humans

This is currently the most promising biomarker. We will measure this biomarker in human urine and a novel MPS IVA rat model. In addition, to increase specificity, we are collaborating with a mass spectrometer manufacturer (SCIEX, Framingham, MA) to establish a method to measure this biomarker by mass spectrometry.

#### **GAGs**

Urinary di-sulfated KS may not be a pharmacodynamic biomarker. Complete data analysis is ongoing.

#### Other biomarkers:

As I showed in the previous review [28], IL-1 $\beta$ , IL-6, IL-18, TNF- $\alpha$ , MMPs may be among the other candidates to measure. We are measuring these biomarkers with the Luminex<sup>TM</sup> xMAP<sup>TM</sup> INTELLIFLEX system by technicians at our institute. The results will be available shortly.

#### References

- 1. Martino, A. T.; Herzog, R. W.; Anegon, I.; Adjali, O. Adeno-Associated Virus, Methods and Protocols. *Methods Mol Biology*, **2011**, *807*, 259–272. https://doi.org/10.1007/978-1-61779-370-7 11.
- 2. Khan, S. A.; Mason, R. W.; Giugliani, R.; Orii, K.; Fukao, T.; Suzuki, Y.; Yamaguchi, S.; Kobayashi, H.; Orii, T.; Tomatsu, S. Glycosaminoglycans Analysis in Blood and Urine of Patients with Mucopolysaccharidosis. *Molecular genetics and metabolism*, **2018**, *125* (1–2), 44–52. https://doi.org/10.1016/j.ymgme.2018.04.011.
- 3. Khan, S. A.; Mason, R. W.; Kobayashi, H.; Yamaguchi, S.; Tomatsu, S. Advances in Glycosaminoglycan Detection. *Molecular genetics and metabolism*, **2020**, *130* (2), 101–109. https://doi.org/10.1016/j.ymgme.2020.03.004.
- 4. Kubaski, F.; Mason, R. W.; Nakatomi, A.; Shintaku, H.; Xie, L.; Vlies, N. N. van; Church, H.; Giugliani, R.; Kobayashi, H.; Yamaguchi, S.; et al. Newborn Screening for Mucopolysaccharidoses: A Pilot Study of Measurement of Glycosaminoglycans by Tandem Mass Spectrometry. *Journal of inherited metabolic disease*, **2017**, *40* (1), 151–158. https://doi.org/10.1007/s10545-016-9981-6.
- 5. Kubaski, F.; Suzuki, Y.; Orii, K.; Giugliani, R.; Church, H. J.; Mason, R. W.; Dung, V. C.; Ngoc, C. T.; Yamaguchi, S.; Kobayashi, H.; et al. Glycosaminoglycan Levels in Dried Blood Spots of Patients with Mucopolysaccharidoses and Mucolipidoses. *Molecular genetics and metabolism*, **2017**, *120* (3), 247–254. https://doi.org/10.1016/j.ymgme.2016.12.010.
- 6. Tomatsu, S.; Shimada, T.; Mason, R. W.; Montano, A. M.; Kelly, J.; LaMarr, W. A.; Kubaski, F.; Giugliani, R.; Guha, A.; Yasuda, E.; et al. Establishment of Glycosaminoglycan Assays for Mucopolysaccharidoses. *Metabolites*, **2014**, *4* (3), 655–679. https://doi.org/10.3390/metabo4030655.
- 7. Hintze, J. P.; Tomatsu, S.; Fujii, T.; Montano, A. M.; Yamaguchi, S.; Suzuki, Y.; Fukushi, M.; Ishimaru, T.; Orii, T. Comparison of Liquid Chromatography-Tandem Mass Spectrometry and Sandwich ELISA for Determination of Keratan Sulfate in Plasma and Urine. *Biomarker insights*, **2011**, *6*, 69–78. https://doi.org/10.4137/bmi.s7451.
- 8. Shimada, T.; Tomatsu, S.; Mason, R. W.; Yasuda, E.; Mackenzie, W. G.; Hossain, J.; Shibata, Y.; Montano, A. M.; Kubaski, F.; Giugliani, R.; et al. Di-Sulfated Keratan Sulfate as a Novel Biomarker for Mucopolysaccharidosis II, IVA, and IVB. *JIMD reports*, **2015**, *21*, 1–13. https://doi.org/10.1007/8904\_2014\_330.
- 9. Tomatsu, S.; Kubaski, F.; Sawamoto, K.; Mason, R. W.; Yasuda, E.; Shimada, T.; Montano, A. M.; Yamaguchi, S.; Suzuki, Y.; Orii, T. Newborn Screening and Diagnosis of Mucopolysaccharidoses: Application of Tandem Mass Spectrometry. *Nihon Masu Sukuriningu Gakkai Shi*, **2014**, *24*, 19–37.
- 10. Hendriksz, C. J.; Burton, B.; Fleming, T. R.; Harmatz, P.; Hughes, D.; Jones, S. A.; Lin, S.; Mengel, E.; Scarpa, M.; Valayannopoulos, V.; et al. Efficacy and Safety of Enzyme Replacement Therapy with BMN 110 (Elosulfase Alfa) for Morquio A Syndrome (Mucopolysaccharidosis IVA): A Phase 3 Randomised Placebocontrolled Study. *J. Inherit. Metab. Dis.*, **2014**, *37* (6), 979–990. https://doi.org/10.1007/s10545-014-9715-6.
- 11. Olney, R. C.; Prickett, T. C. R.; Espiner, E. A.; Mackenzie, W. G.; Duker, A. L.; Ditro, C.; Zabel, B.; Hasegawa, T.; Kitoh, H.; Aylsworth, A. S.; et al. C-Type Natriuretic Peptide Plasma Levels Are Elevated in Subjects With Achondroplasia, Hypochondroplasia, and Thanatophoric Dysplasia. *J Clin Endocrinol Metabolism*, **2015**, *100* (2), E355–E359. https://doi.org/10.1210/jc.2014-2814.

- 12. Klag, K. A.; Horton, W. A. Advances in Treatment of Achondroplasia and Osteoarthritis. *Hum. Mol. Genet.*, **2016**, *25* (R1), R2–R8. https://doi.org/10.1093/hmg/ddv419.
- 13. Franceschi, L. D.; Roseti, L.; Desando, G.; Facchini, A.; Grigolo, B. A Molecular and Histological Characterization of Cartilage from Patients with Morquio Syndrome. *Osteoarthr Cartilage*, **2007**, *15* (11), 1311–1317. https://doi.org/10.1016/j.joca.2007.04.008.
- 14. Dvorak-Ewell, M.; Wendt, D.; Hague, C.; Christianson, T.; Koppaka, V.; Crippen, D.; Kakkis, E.; Vellard, M. Enzyme Replacement in a Human Model of Mucopolysaccharidosis IVA In Vitro and Its Biodistribution in the Cartilage of Wild Type Mice. *PLoS ONE*, **2010**, *5* (8), e12194. https://doi.org/10.1371/journal.pone.0012194.
- 15. Álvarez, J. Victor.; Bravo, S. B.; Chantada-Vázquez, M. P.; Pena, C.; Colón, C.; Tomatsu, S.; Otero-Espinar, F. J.; Couce, M. L. Morquio A Syndrome: Identification of Differential Patterns of Molecular Pathway Interactions in Bone Lesions. *Int. J. Mol. Sci.*, **2024**, *25* (6), 3232. https://doi.org/10.3390/ijms25063232.
- 16. Sorokina, L. V.; Shahbazian-Yassar, R.; Shokuhfar, T. Collagen Biomineralization: Pathways, Mechanisms, and Thermodynamics. *Emergent Mater.*, **2021**, *4* (5), 1205–1224. https://doi.org/10.1007/s42247-021-00226-1.
- 17. Bakkalci, D.; Micalet, A.; Hosni, R. A.; Moeendarbary, E.; Cheema, U. Associated Changes in Stiffness of Collagen Scaffolds during Osteoblast Mineralisation and Bone Formation. *BMC Res. Notes*, **2022**, *15* (1), 310. https://doi.org/10.1186/s13104-022-06203-z.
- 18. Garnero, P. The Role of Collagen Organization on the Properties of Bone. *Calcif. Tissue Int.*, **2015**, 97 (3), 229–240. https://doi.org/10.1007/s00223-015-9996-2.
- 19. Conrozier, T.; Ferrand, F.; Poole, A. R.; Verret, C.; Mathieu, P.; Ionescu, M.; Vincent, F.; Piperno, M.; Spiegel, A.; Vignon, E. Differences in Biomarkers of Type II Collagen in Atrophic and Hypertrophic Osteoarthritis of the Hip: Implications for the Differing Pathobiologies. *Osteoarthr. Cartil.*, **2007**, *15* (4), 462–467. https://doi.org/10.1016/j.joca.2006.09.002.
- 20. Arunrukthavon, P.; Heebthamai, D.; Benchasiriluck, P.; Chaluay, S.; Chotanaphuti, T.; Khuangsirikul, S. Can Urinary CTX-II Be a Biomarker for Knee Osteoarthritis? *Arthroplasty*, **2020**, *2* (1), 6. https://doi.org/10.1186/s42836-020-0024-2.
- 21. Cheng, H.; Hao, B.; Sun, J.; Yin, M. C-Terminal Cross-Linked Telopeptides of Type II Collagen as Biomarker for Radiological Knee Osteoarthritis: A Meta-Analysis. *CARTILAGE*, **2020**, *11* (4), 512–520. https://doi.org/10.1177/1947603518798884.
- 22. Nicolini, A.; Mansur, N.; Dreyfuss, J.; Ejnisman, B.; Cohen, M.; Astur, D. Avaliação Do Biomarcador CTX-II Em Pacientes Com Ruptura Do Ligamento Cruzado Anterior: Estudo Piloto\*. *Rev. Bras. Ortop.*, **2020**, *56* (03), 326–332. https://doi.org/10.1055/s-0040-1712139.
- 23. Song, Q. Q.; Sun, L. Y.; Li, C. H.; Liu, Y. J.; Cui, S. L.; Liu, Y. Q.; Cao, Y. H.; Pei, J. R.; Wang, Y.; Lian, W.; et al. The Urinary Levels of CTX-II, C2C, PYD, and Helix-II Increased among Adults with KBD: A Cross-Sectional Study. *J. Orthop. Surg. Res.*, **2019**, *14* (1), 328. https://doi.org/10.1186/s13018-019-1392-6.
- 24. Cahue, S.; Sharma, L.; Dunlop, D.; Ionescu, M.; Song, J.; Lobanok, T.; King, L.; Poole, A. R. The Ratio of Type II Collagen Breakdown to Synthesis and Its Relationship with the Progression of Knee Osteoarthritis. *Osteoarthr. Cartil.*, **2007**, *15* (7), 819–823. https://doi.org/10.1016/j.joca.2007.01.016.
- 25. Conrozier, T.; Poole, A. R.; Ferrand, F.; Mathieu, P.; Vincent, F.; Piperno, M.; Verret, C.; Ionescu, M.; Vignon, E. Serum Concentrations of Type II Collagen Biomarkers (C2C, C1, 2C and CPII) Suggest Different Pathophysiologies in Patients with Hip Osteoarthritis. *Clin. Exp. Rheumatol.*, **2008**, *26* (3), 430–435.

- 26. Mullan, R. H.; Matthews, C.; Bresnihan, B.; FitzGerald, O.; King, L.; Poole, A. R.; Fearon, U.; Veale, D. J. Early Changes in Serum Type Ii Collagen Biomarkers Predict Radiographic Progression at One Year in Inflammatory Arthritis Patients after Biologic Therapy. *Arthritis Rheum.*, **2007**, *56* (9), 2919–2928. https://doi.org/10.1002/art.22843.
- 27. Bay-Jensen, A.-C.; Tabassi, N. C.; Sondergaard, L. V.; Andersen, T. L.; Dagnaes-Hansen, F.; Garnero, P.; Kassem, M.; Delaissé, J.-M. The Response to Oestrogen Deprivation of the Cartilage Collagen Degradation Marker, CTX-II, Is Unique Compared with Other Markers of Collagen Turnover. *Arthritis Res. Ther.*, **2009**, *11* (1), R9. https://doi.org/10.1186/ar2596.
- 28. Ago, Y.; Rintz, E.; Musini, K. S.; Ma, Z.; Tomatsu, S. Molecular Mechanisms in Pathophysiology of Mucopolysaccharidosis and Prospects for Innovative Therapy. *Int. J. Mol. Sci.*, **2024**, *25* (2), 1113. https://doi.org/10.3390/ijms25021113.
- 29. Doherty, C.; Stapleton, M.; Piechnik, M.; Mason, R. W.; Mackenzie, W. G.; Yamaguchi, S.; Kobayashi, H.; Suzuki, Y.; Tomatsu, S. Effect of Enzyme Replacement Therapy on the Growth of Patients with Morquio A. *J. Hum. Genet.*, **2019**, *64* (7), 625–635. https://doi.org/10.1038/s10038-019-0604-6.
- 30. Olney, R. C.; Permuy, J. W.; Prickett, T. C. R.; Han, J. C.; Espiner, E. A. Amino-terminal Propeptide of C-type Natriuretic Peptide (NTproCNP) Predicts Height Velocity in Healthy Children. *Clin. Endocrinol.*, **2012**, 77 (3), 416–422. https://doi.org/10.1111/j.1365-2265.2012.04392.x.

### Discussion Unmet goals

#### Aim 1.

We have reached our goal of over 60 actively enrolled participants and will continue to have follow-up visits as they are interested.

- 1. We will not have enough to achieve 4 visits; therefore, we will resubmit the grant based on the achievements.
- 2. We will summarize the data and will publish each test data.

#### Aim 2.

- 1. We will continue to assay the biomarkers, including glycosaminoglycans (C6S and KS), Collagen, and Inflammatory factors.
- 2. We will submit the manuscripts with data of biological biomarkers.

#### **PUBLICATIONS** (other achievements)

#### 2022

- Poletto E, Colella P, Pimentel Vera LN, Khan S, **Tomatsu S**, Baldo G, Gomez-Ospina N. Improved engraftment and therapeutic efficacy by human genome-edited hematopoietic stem cells with Busulfan-based myeloablation. Mol Ther Methods Clin Dev. 2022 Apr 19;25:392-409. doi: 10.1016/j.omtm.2022.04.009. PMID: 35573043; PMCID: PMC9065050.
- Rintz E, Węgrzyn G, Fujii T, **Tomatsu S**. Molecular Mechanism of Induction of Bone Growth by the C-Type Natriuretic Peptide. Int J Mol Sci. 2022 May 25;23(11):5916. doi: 10.3390/ijms23115916. PMID: 35682595; PMCID: PMC9180634.
- Leal AF, Fnu N, Benincore-Flórez E, Herreño-Pachón AM, Echeverri-Peña OY, Alméciga-Díaz CJ, **Tomatsu S**. The landscape of CRISPR/Cas9 for inborn errors of metabolism. Mol Genet Metab. 2023 Jan;138(1):106968. doi: 10.1016/j.ymgme.2022.106968. Epub 2022 Dec 7. PMID: 36525790; PMCID: PMC10199355.
- Jalal K, Carter RL, Barczykowski A, **Tomatsu S**, Langan TJ. A Roadmap for Potential Improvement of Newborn Screening for Inherited Metabolic Diseases Following Recent Developments and Successful Applications of Bivariate Normal Limits for Pre-Symptomatic Detection of MPS I, Pompe Disease, and Krabbe Disease.

- Int J Neonatal Screen. 2022 Nov 15;8(4):61. doi: 10.3390/ijns8040061. PMID: 36412587; PMCID: PMC9680456.
- Celik B, Cicek K, Leal AF, **Tomatsu S**. Regulation of Molecular Targets in Osteosarcoma Treatment. Int J Mol Sci. 2022 Oct 20;23(20):12583. doi: 10.3390/ijms232012583. PMID: 36293439; PMCID: PMC9604206.
- Piechnik M, Amendum PC, Sawamoto K, Stapleton M, Khan S, Fnu N, Álvarez V, Pachon AMH, Danos O, Bruder JT, Karumuthil-Melethil S, **Tomatsu S**. Sex Difference Leads to Differential Gene Expression Patterns and Therapeutic Efficacy in Mucopolysaccharidosis IVA Murine Model Receiving AAV8 Gene Therapy. Int J Mol Sci. 2022 Oct 21;23(20):12693. doi: 10.3390/ijms232012693. PMID: 36293546; PMCID: PMC9604118.
- Pan X, Taherzadeh M, Bose P, Heon-Roberts R, Nguyen ALA, Xu T, Pará C, Yamanaka Y, Priestman DA, Platt FM, Khan S, Fnu N, **Tomatsu S**, Morales CR, Pshezhetsky AV. Glucosamine amends CNS pathology in mucopolysaccharidosis IIIC mouse expressing misfolded HGSNAT. J Exp Med. 2022 Aug 1;219(8):e20211860. doi: 10.1084/jem.20211860. Epub 2022 Jun 15. PMID: 35704026; PMCID: PMC9204472.
- Rintz E, Higuchi T, Kobayashi H, Galileo DS, Wegrzyn G, **Tomatsu S**. Promoter considerations in the design of lentiviral vectors for use in treating lysosomal storage diseases. Mol Ther Methods Clin Dev. 2021 Nov 24;24:71-87. doi: 10.1016/j.omtm.2021.11.007. PMID: 34977274; PMCID: PMC8688940.

#### 2023

- Leal AF, Fnu N, Benincore-Flórez E, Herreño-Pachón AM, Echeverri-Peña OY, Alméciga-Díaz CJ, **Tomatsu S**. The landscape of CRISPR/Cas9 for inborn errors of metabolism. Mol Genet Metab. 2023 Jan;138(1):106968. doi: 10.1016/j.ymgme.2022.106968. Epub 2022 Dec 7. PMID: 36525790; PMCID: PMC10199355.
- Khan SA, Nidhi FNU, Amendum PC, **Tomatsu S**. Detection of Glycosaminoglycans in Biological Specimens. Methods Mol Biol. 2023;2619:3-24. doi: 10.1007/978-1-0716-2946-8\_1. PMID: 36662458; PMCID: PMC10199356.
- Rintz E, Herreño-Pachón AM, Celik B, Nidhi F, Khan S, Benincore-Flórez E, **Tomatsu S**. Bone Growth Induction in Mucopolysaccharidosis IVA Mouse. Int J Mol Sci. 2023 Jun 8;24(12):9890. doi: 10.3390/ijms24129890. PMID: 37373036; PMCID: PMC10298227.
- Theroux MC, DiCindio S, Averill LW, Pizarro C, Oommen A, Bober MB, Ditro C, Campbell J, Duker AL, Jones T, Passi V, Barth P, Schmidt RJ, Little M, Mackenzie S, **Tomatsu S**, Mackenzie WG. Tracheal Narrowing and Its Impact on Anesthesia Care in Patients With Morquio A (Mucopolysaccharidosis Type IVA): An Observational Study. Anesth Analg. 2023 Nov 1;137(5):1075-1083. doi: 10.1213/ANE.000000000006513. Epub 2023 May 9. PMID: 37862598; PMCID: PMC10634225.
- Leal AF, Celik B, Fnu N, Khan S, **Tomatsu S**, Alméciga-Díaz CJ. Iron oxide-coupled CRISPR-nCas9-based genome editing assessment in mucopolysaccharidosis IVA mice. Mol Ther Methods Clin Dev. 2023 Nov 7;31:101153. doi: 10.1016/j.omtm.2023.101153. PMID: 38107675; PMCID: PMC10724691.
- Leal AF, Alméciga-Díaz CJ, **Tomatsu S**. Mucopolysaccharidosis IVA: Current Disease Models and Drawbacks. Int J Mol Sci. 2023 Nov 9;24(22):16148. doi: 10.3390/ijms242216148. PMID: 38003337; PMCID: PMC10671113.

#### 2024

- Ago Y, Rintz E, Musini KS, Ma Z, Tomatsu S. Molecular Mechanisms in Pathophysiology of Mucopolysaccharidosis and Prospects for Innovative Therapy. Int J Mol Sci. 2024 Jan 17;25(2):1113. doi: 10.3390/ijms25021113.PMID: 38256186.
- Khan SA, Nidhi F, Leal AF, Celik B, Herreño-Pachón AM, Saikia S, Benincore-Flórez E, Ago Y, Tomatsu S. Glycosaminoglycans in mucopolysaccharidoses and other disorders. Adv Clin Chem. 2024;122:1-52. doi: 10.1016/bs.acc.2024.06.011. Epub 2024 Jul 23. PMID: 39111960.
- Leal AF, Herreno-Pachón AM, Benincore-Flórez E, Karunathilaka A, Tomatsu S. Current Strategies for Increasing Knock-In Efficiency in CRISPR/Cas9-Based Approaches. Int J Mol Sci. 2024 Feb 20;25(5):2456. doi: 10.3390/ijms25052456.
- Álvarez JV, Bravo SB, Chantada-Vázquez MP, Pena C, Colón C, **Tomatsu S**, Otero-Espinar FJ, Couce ML. Morquio A Syndrome: Identification of Differential Patterns of Molecular Pathway Interactions in Bone Lesions. Int J Mol Sci. 2024 Mar 12;25(6):3232. doi: 10.3390/ijms25063232.PMID: 38542208
- Rintz E, Celik B, Fnu N, Herreño-Pachón AM, Khan S, Benincore-Flórez E, **Tomatsu S**. Adeno-associated virus-based gene therapy delivering combinations of two growth-associated genes to MPS IVA mice. Mol Ther Nucleic Acids. 2024 May 7;35(2):102211. doi: 10.1016/j.omtn.2024.102211. eCollection 2024 Jun 11. PMID: 38831899.

- Bradford A, Klipner K, Mackenzie WSG, **Tomatsu S**. Accelerating Medicines Partnership Bespoke Gene Therapy Consortium for Rare Disorders. Nippon Rynshou. 2024 May 82;5 769-777.Celik B, Leal AF, **Tomatsu S**. Potential Targeting Mechanisms for Bone-Directed Therapies. Int J Mol Sci. 2024, *25*(15), 8339; https://doi.org/10.3390/ijms25158339.
- Celik B, Rintz E, Sansanwal N, Khan S, Bigger B, **Tomatsu S**. Lentiviral Vector-Mediated Ex Vivo Hematopoietic Stem Cell Gene Therapy for MPS IVA Murine Model. Hum Gene Ther. 2024 Oct 24. doi: 10.1089/hum.2024.094.
- Herreño-Pachón AM, Sawamoto K, Stapleton M, Khan S, Piechnik M, J. Álvarez V, **Tomatsu S**. AAV Gene Transfer Ameliorates the Progression of Skeletal Lesions in Mucopolysaccharidosis IVA Mice. Hum Gene Ther. 2024 Oct 25. doi: 10.1089/hum.2024.096.

#### 2025

- Khan S, Ago Y, **Tomatsu S**. VIEWPOINT: AAV gene therapy for rare disorders: generate critical data on safety and efficacy. Med (accepted).
- Khan SA, Álvarez JA, Nidhi F, Florez EB, **Tomatsu S**. Evaluation of AAV vectors with tissue-specific or ubiquitous promoters in a mouse model of mucopolysaccharidosis type IVA. Mol Ther Methods Clin Dev. (accepted).

# Supplementary Table 1 (3/11/2025)

| Study<br>ID | Sex | Age (Years) at<br>Enrollment | Race | Ethnicity |
|---|---|---|---|---|
| M01 | F | 17 | White or Caucasian | Non-Hispanic or Latino |
| M02 | F | 38 | Asian | Non-Hispanic or Latino |
| M03 | F | 24 | White or Caucasian | Non-Hispanic or Latino |
| M04 | F | 42 | White or Caucasian | Non-Hispanic or Latino |
| M05 | F | 18 | White or Caucasian | Non-Hispanic or Latino |
| M06 | F | 19 | White or Caucasian | Non-Hispanic or Latino |
| M07 | М | 32 | White or Caucasian | Non-Hispanic or Latino |
| M08 | М | 8 | White or Caucasian | Hispanic or Latino |
| M10 | М | 10 | White or Caucasian | Non-Hispanic or Latino |
| M11 | F | 14 | White or Caucasian | Non-Hispanic or Latino |
| M12 | F | 26 | White or Caucasian | Non-Hispanic or Latino |
| M13 | М | 12 | Black or African American | Non-Hispanic or Latino |
| M14 | F | 16 | White or Caucasian | Hispanic or Latino |
| M15 | М | 5 | White or Caucasian | Non-Hispanic or Latino |
| M16 | М | 5 | Multiple Races | Non-Hispanic or Latino |
| M19 | F | 9 | Black or African American | Non-Hispanic or Latino |
| M20 | F | 9 | White or Caucasian | Non-Hispanic or Latino |
| M21 | М | 5 | White or Caucasian | Non-Hispanic or Latino |
| M22 | М | 8 | White or Caucasian | Non-Hispanic or Latino |
| M25 | М | 41 | White or Caucasian | Non-Hispanic or Latino |
| M26 | М | 11 | Multiple Races | Hispanic or Latino |
| M27 | М | 9 | White or Caucasian | Hispanic or Latino |
| M28 | F | 30 | Multiple Races | Non-Hispanic or Latino |
| M30 | F | 43 | White or Caucasian | Non-Hispanic or Latino |
| M31 | М | 9 | Black or African American | Non-Hispanic or Latino |
| M32 | F | 45 | White or Caucasian | Non-Hispanic or Latino |
| M33 | F | 29 | White or Caucasian | Non-Hispanic or Latino |
| M34 | М | 27 | White or Caucasian | Non-Hispanic or Latino |
| M35 | М | 11 | Other | Hispanic or Latino |
| M36 | F | 25 | Other | Non-Hispanic or Latino |
| M37 | М | 18 | Other | Non-Hispanic or Latino |
| M41 | М | 35 | White or Caucasian | Non-Hispanic or Latino |
| M42 | F | 27 | White or Caucasian | Non-Hispanic or Latino |
| M43 | M | 28 | White or Caucasian | Non-Hispanic or Latino |
| M44 | F | 23 | White or Caucasian | Non-Hispanic or Latino |
| M45 | F | 60 | White or Caucasian | Non-Hispanic or Latino |
| M46 | F | 6 | White or Caucasian | Hispanic or Latino |
| M47 | F | 23 | White or Caucasian | Hispanic or Latino |
| M48 | F | 12 | White or Caucasian | Hispanic or Latino |
| M49 | M | 6 | White or Caucasian | Hispanic or Latino |
| M50 | F | 4 | White or Caucasian | Non-Hispanic or Latino |
| M51 | M | 2 | White or Caucasian | Non-Hispanic or Latino |
| M52 | F | 3 | Multiple Races | Hispanic or Latino |
| M53 | F | 22 | Asian | Non-Hispanic or Latino |
| M54 | F | 35 | White or Caucasian | Non-Hispanic or Latino |
| M55 | F | 4 | White or Caucasian | Non-Hispanic or Latino |
| M56 | F | 3 | White or Caucasian | Non-Hispanic or Latino |
| M57 | М | 10 months | White or Caucasian | Non-Hispanic or Latino |
| M58 | M | 6 | White or Caucasian | Non-Hispanic or Latino |
| M59 | M | 5 | White or Caucasian | Non-Hispanic or Latino |

| M60 | F | 25 | Other | Hispanic or Latino |
|-----|---|-----------|--------------------|------------------------|
| M63 | H | 22 | White or Caucasian | Non-Hispanic or Latino |
| M64 | М | 5 | Multiple Races | Non-Hispanic or Latino |
| M65 | М | 6 | Multiple Races | Non-Hispanic or Latino |
| M66 | H | 3 | White or Caucasian | Hispanic or Latino |
| M67 | М | 11 | White or Caucasian | Non-Hispanic or Latino |
| M68 | М | 45 | White or Caucasian | Hispanic or Latino |
| M69 | М | 2 | Asian | Non-Hispanic or Latino |
| M70 | M | 13 | White or Caucasian | Non-Hispanic or Latino |
| M71 | М | 8 | White or Caucasian | Non-Hispanic or Latino |
| M72 | М | 2 | Asian | Hispanic or Latino |
| M73 | F | 3 | White or Caucasian | Non-Hispanic or Latino |
| M74 | F | 37 | White or Caucasian | Non-Hispanic or Latino |
| M76 | F | 10 months | White or Caucasian | Non-Hispanic or Latino |
| M77 | F | 2 | White or Caucasian | Non-Hispanic or Latino |
| M78 | М | 11 | White or Caucasian | Non-Hispanic or Latino |

### Supplementary Table 2 (3/11/2025)

| Estimated Number of Actively Enrolled Participants to Complete Each Study Visit Before May 2026 | |
|---|---|
| Baseline | 66 |
| 18 months | 62 |
| 36 months | 50 |
| 54 months | 0 |

#### ClinicalTrials.gov Protocol Registration and Results System (PRS)

750932-25 NCT05284006 Non-invasive Functional Assessment and Pathogenesis of Morquio A (NIFAMA)

NIH: <u>Study Record | Beta ClinicalTrials.gov</u> Clinicaltrials.gov: <u>Non-invasive Functional Assessment and Pathogenesis of Morquio A - Full Text View -</u> ClinicalTrials.gov

# Describe briefly what you plan to do during the next reporting period to accomplish the goals and objectives.

We have reached our goal of over 60 actively enrolled participants and will continue to have follow-up visits as they are interested.

- 1. We will not have enough to achieve 4 visits because of the initial delay due to COVID19 pandemic. We will accommodate the patients as much as possible to increase the number of visits in total. We will also resubmit the grant to accomplish 4 visits.
- 2. We will summarize the data and will publish each test data in the 5<sup>th</sup> year period.
- 3. We will continue to assay the biomarkers, including glycosaminoglycans (C6S and KS), Nt-pro-CNP, Collagen, and Inflammatory factor and will correlate these biological biomarkers with the clinical phenotype, especially skeletal symptoms. We will submit the manuscripts with data of biological biomarkers.

Include any important modifications to the original plans. Provide a scientific justification for any changes involving research with human subjects or vertebrate animals. A detailed description of such changes must be provided under Changes.